CLINICAL TRIAL: NCT03873181
Title: Post-Market Evaluation of HEMOBLAST™ Bellows Performance and Safety in Laparoscopic Abdominal, Gynecological and Urological Surgery
Brief Title: Post-Market Evaluation of HEMOBLAST™ Bellows in Laparoscopic Abdominal, Gynecological, and Urological Surgery
Acronym: NOBLE-Laparo
Status: Completed | Type: Observational
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ETC 2018-002
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Hemostasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: HEMOBLAST™ Bellows — Surgeon has chosen to use HEMOBLAST™ Bellows as an adjunct to hemostasis when control of minimal, mild, or moderate bleeding by conventional procedures is ineffective or impractical in laparoscopic abdominal, gynecological, or urological surgeries.

SUMMARY:
A prospective, multi-center, multi-national single arm study to evaluate the performance and safety of HEMOBLAST™ Bellows in laparoscopic abdominal, gynecological, and urological surgery.

DETAILED DESCRIPTION:
A prospective, multi-center, multi-national single arm study conducted in Austria, France, and Germany to evaluate the performance and safety of HEMOBLAST™ Bellows in laparoscopic abdominal, gynecological, and urological surgery. Up to 100 subjects will be enrolled at up to 10 sites, with a minimum of 8 subjects enrolled in each surgical specialty.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Patient is undergoing a non-emergent laparoscopic abdominal, gynecological, or urological surgery
* Patient is willing and able to give prior written informed consent for investigation participation;
* Patient is 18 years of age or older.

Intra-operative Inclusion Criteria

* Patient has one or more target bleeding sites (TBS) for which control of bleeding by conventional procedures is ineffective or impractical.
* The TBS(s) has been treated with HEMOBLAST™ Bellows and the HEMOBLAST™ Bellows Laparoscopic Applicator as per their instructions for use.

Exclusion Criteria:

* Patient is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding;
* Patient has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
* Patient has religious or other objections to porcine, bovine, or human components;
* Patient has any significant coagulation disorder;
* Patient has any other contraindications, warnings, precautions of the Approved Instruction For Use of HEMOBLAST™ Bellows preventing his/ her inclusion
* Patient is not appropriate for inclusion in the clinical trial, per the medical opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing laparoscopic abdominal, gynecological, or urological procedures that meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Achievement of Hemostasis | Intraoperatively, expected within 3-10 minutes of application
  The proportion of subjects for which hemostasis was achieved after application of HEMOBLAST™ Bellows.

SECONDARY OUTCOMES:
Re-bleeding at Target Bleeding Site | Intraoperative, prior to surgical closure of the subject
  The rate of target bleeding site re-bleeding after hemostasis has been achieved with HEMOBLAST™ Bellows
Re-operation due to bleeding | Post-operatively, expected within 1-30 days of the surgical procedure
  The rate of re-operation due to post-operative bleeding/hemorrhage after treatment with HEMOBLAST™ Bellows

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vilz, MD, Principal Investigator — University Hospital, Bonn
Locations (8):
- University Hospital Salzburg, Salzburg, Austria
- France (3):
  - Hôpital Beaujon, Clichy
  - CHU Grenoble, Grenoble
  - Hôpital Saint Jospeh, Paris
- Germany (4):
  - University Hospital Bonn, Bonn
  - Kliniken der Stadt Koln, Krankenhaus Merheim, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Asklepios Klinik Barmbek, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided